CLINICAL TRIAL: NCT00155909
Title: To Investigate Risk Factors of Radiation Pneumonitis, Fibrosis, and Impairment of Quality of Life by Radiotherapeutic Dosimetric and Biological Parameters for Lung Cancer Patients Receiving Thoracic Radiotherapy
Brief Title: Risk Factors of Radiation Pneumonitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261700803; NTUH-92N013
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2005-06

CONDITIONS: Radiation Pneumonitis
Keywords: Radiation Pneumonitis; Radiotherapy Planning, Computer-Assisted
MeSH Terms: conditions — Radiation Pneumonitis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
A prospective observational study to evaluate clinical, dosimetrical, functional, and biological factors in predicting radiation pneumonitis.

DETAILED DESCRIPTION:
We propose a prospective observational study to investigate the combinational effect of radiotherapeutic dosimetric parameters [mean lung dose & percentage of lung volume receiving at least 20Gy (V20)] and biological parameters [interleukin-6(IL6) & transforming growth factor beta (TGFB)] in predicting radiation pneumonitis, fibrosis, and change of QoL among at least fifty-three lung cancer patients. Eligibility included pathological or cytological proven small cell or non small cell lung cancer, thoracic RT planned for more than 30Gy [if fraction size >= 3Gy/fx] or 40Gy [if fraction size < 3 Gy/Fx], ECOG performance status [PS] 0-2, body weight loss [BWL] <=10% in previous 6 months, no prior thoracic RT and signed informed consent prior to study entry. Basic pre-radiotherapy information will be collected, which included BWL, ECOG PS, AJCC stage [I-IV], primary lesion site, history of smoking/coexisting lung disease/dosage of chemotherapy/surgical resection, albumin level, and pulmonary function test of FEV1/VC/DLCO(optional). Computed tomography [CT] of the whole lung in treatment position with reference mark will be done for calculation of V20 and mean lung dose. Blood test of IL6, TGFB by ELISA will be done before and after RT after storage at -80℃. Bronchial-alveolar lavage test of IL6, TGFB by ELISA will be done before and after RT if clinical available. Self-reported questionnaire [EORTC C30 & L13] will be collected before and after RT and in every follow up visits after double-checked by trained assistants. RT must be given by photon energies >=6MV. Radiation pneumonitis and fibrosis will be assessed according to common toxicity criteria 3 [CTC-3] weekly during RT and in every follow up visits. Chi-square test, logistic regression, and proportional hazard ratio method will be used to investigate whether the parameter(s) can be effective in predicting radiation related sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adults (age >=20 y/o)
* Pathological or cytological proven small cell or non small cell lung cancer
* Thoracic RT planned for more than 30Gy [if fraction size >= 3Gy/fx] or 40Gy [if fraction size < 3 Gy/Fx]
* ECOG PS 0-2
* Body weight loss <=10% in previous 6 months

Exclusion Criteria:

* prior thoracic RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53
Dates: Start 2003-07; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ru Chien, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan